CLINICAL TRIAL: NCT02338609
Title: Long-term Follow-up Study to Monitor the Growth and Development of Pediatric Patients Previously Treated With Everolimus in Study CRAD001M2301 (EXIST-LT)
Brief Title: Long-term Monitoring of Growth and Development of Pediatric Patients Previously Treated With Everolimus
Acronym: EXIST-LT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRAD001M2305; 2013-003795-13 (EudraCT Number)
Record Dates: First submitted 2014-12-01; First posted 2015-01-14 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Growth and Development
Keywords: TSC-associated SEGA,; height,; weight,; Tanner Stage,; growth development,; everolimus,; RAD001
MeSH Terms: conditions — Body Weight | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental): All patients will have been previously treated with everolimus as part of CRAD001M2301. Continued treatment with everolimus is allowed but not required for participation in this study.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — At the discretion of the investigator, pediatric patients could be treated with commercially available everolimus, as per local product information / standard of care. Treatment duration and dose modifications were at the investigator's discretion, as per the local product information.

SUMMARY:
The primary objective of CRAD001M2305 was to report the long-term effects of everolimus treatment on height, weight and sexual development (using Tanner Stages) in children and adolescents with Tuberous Sclerosis Complex (TSC)-associated with Subependymal Giant Cell Astrocytoma (SEGA). The study monitored the growth and development of pediatric patients with TSC-associated SEGA, previously enrolled in CRAD001M2301 (NCT00789828) until they reach Tanner Stage V, or until age 16 for females or 17 for males whichever occurred first.

DETAILED DESCRIPTION:
CRAD001M2305 was a prospective, multi-center phase IIIb/IV study. This study investigated if the physical and sexual development of pediatric patients was affected by previous or ongoing treatment with everolimus. The study monitored the growth and development of pediatric patients with TSC-associated SEGA, previously enrolled in CRAD001M2301(NCT00789828) until they reached Tanner Stage V, or until age 16 for females or 17 for males whichever occurred first. Continued treatment with everolimus was at investigator discretion and was not required for participation in CRAD001M2305. Growth (height, weight), and sexual development (Tanner Stages, sex hormone levels, age at menarche, thelarche (females) and adrenarche (males)), and brain development (assessed by TAND Checklist, dates of brain MRI) of patients participating in this long-term follow-up study was followed at annual visits to the site until patients achieve Tanner Stage V or age 16 (females), age 17 (males) whichever occurred first. Adverse events, concomitant medication, appearance of menarche, were monitored and data collected every 3 months ("3-monthly"). Unless clinically indicated these 3-monthly visits were performed per telephone.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric female patients who were on study treatment in study [CRAD001M2301] within the past 6 months and have not reached Tanner Stage V or age 16 at the time of completion of [CRAD001M2301] or
* Pediatric male patients who were on study treatment in study [CRAD001M2301] within the past 6 months and have not reached Tanner Stage V or age 17 at the time of completion of [CRAD001M2301]
* Written informed consent according to local guidelines

Exclusion Criteria:

* Pediatric female patients who were on study treatment in CRAD001M2301 and have not reached Tanner Stage V but are within 3 month of turning age 16 or
* Pediatric male patients who were on study treatment in CRAD001M2301 and have not reached Tanner Stage V but are within 3 months of turning age 17
* Any patient who was pregnant prior to start of CRAD001M2305

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (4):
  - University Of California LA SC, Los Angeles, California
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - Cinn Children Hosp Medical Center SC, Cincinnati, Ohio
  - Texas Scottish Rite Hos for Child SC, Dallas, Texas
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 6 investigative sites in 3 countries.
Pre-assignment Details: All the pediatric patients enrolled into the current study had been treated with everolimus in the parent study CRAD001M2301.
Groups:
- Everolimus: Participants were treated with everolimus as part of CRAD001M2301. Continued treatment with everolimus is allowed but not required for participation in this study.
Period: Overall Study
Arm/Group | Everolimus
Started | 15
Safety Analysis Set (All pediatric participants enrolled in this study who had at least one-post baseline safety assessment.) | 14
Completed | 13
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.390 (3.5647)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1
  Caucasian | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Tanner Stage V at or Before Age 16 (Females) or 17 (Males)
Description: Tanner Staging, also known as Sexual Maturity Rating (SMR), is an objective classification system that providers use to document and track the development and sequence of secondary sex characteristics of children during puberty. Tanner Stage included two components for boys (testis and pubic hair) and two components for girls (breast development and pubic hair).
  Tanner Stage V:
  Males and females: Terminal hair that extends beyond the inguinal crease onto the thigh.
  Female Breast Development Scale: Areolar mound recedes into single breast contour with areolar hyperpigmentation, papillae development, and nipple protrusion.
  Male External Genitalia Scale: > 20 ml (or > 4.5 cm long)
Time Frame: Annually, up to 14 years from the first visit in parent study CRAD001M2301 (including up to 9 years of follow-up in study CRAD001M2305)
Population: The Full Analysis Set for sexual development (FAS Puberty) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Female: number analyzed (Participants) | 8
  Female | 4
  Male: number analyzed (Participants) | 7
  Male | 6

2. Primary Outcome: Number of Participants With Notably Low and Notably High Height and Body Mass Index (BMI) Standard Deviation Score (SDS)
Description: Height and body weight (with minimal clothing, without shoes) were measured annually. The height standard deviation score (SDS) and BMI SDS were calculated based on height/BMI data collected during the study and published reference height/BMI information (De Onis M, et al. Development of a WHO growth reference for school-aged children and adolescents. Bull World Health Organ. 2007 Sep;85(9):660-7). The number of participants with height and BMI SDS values lower than the 5th percentile (notably low) or higher than the 95th percentile (notably high) are reported.
  The baseline corresponds to the last available assessment on or before the start of everolimus in the parent study CRAD001M2301. The assessment is performed up to age of 12 years.
Time Frame: Baseline, annually up to Year 10 of treatment since the start of everolimus in parent study CRAD001M2301 (including a median of 5 years of exposure to everolimus in study CRAD001M2305)
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Height SDS-notably low-Baseline | 2
  Height SDS-notably low-Year 1 | 1
  Height SDS-notably low-Year 2: number analyzed (Participants) | 14
  Height SDS-notably low-Year 2 | 2
  Height SDS-notably low-Year 3 | 2
  Height SDS-notably low-Year 4 | 2
  Height SDS-notably low-Year 5: number analyzed (Participants) | 12
  Height SDS-notably low-Year 5 | 2
  Height SDS-notably low-Year 6: number analyzed (Participants) | 12
  Height SDS-notably low-Year 6 | 1
  Height SDS-notably low-Year 7: number analyzed (Participants) | 9
  Height SDS-notably low-Year 7 | 1
  Height SDS-notably low-Year 8: number analyzed (Participants) | 9
  Height SDS-notably low-Year 8 | 0
  Height SDS-notably low-Year 9: number analyzed (Participants) | 8
  Height SDS-notably low-Year 9 | 0
  Height SDS-notably low-Year 10: number analyzed (Participants) | 3
  Height SDS-notably low-Year 10 | 0
  Height SDS-notably high-Baseline | 1
  Height SDS-notably high-Year 1 | 0
  Height SDS-notably high-Year 2: number analyzed (Participants) | 14
  Height SDS-notably high-Year 2 | 0
  Height SDS-notably high-Year 3 | 0
  Height SDS-notably high-Year 4 | 1
  Height SDS-notably high-Year 5: number analyzed (Participants) | 12
  Height SDS-notably high-Year 5 | 0
  Height SDS-notably high-Year 6: number analyzed (Participants) | 12
  Height SDS-notably high-Year 6 | 1
  Height SDS-notably high-Year 7: number analyzed (Participants) | 9
  Height SDS-notably high-Year 7 | 1
  Height SDS-notably high-Year 8: number analyzed (Participants) | 9
  Height SDS-notably high-Year 8 | 1
  Height SDS-notably high-Year 9: number analyzed (Participants) | 8
  Height SDS-notably high-Year 9 | 0
  Height SDS-notably high-Year 10: number analyzed (Participants) | 3
  Height SDS-notably high-Year 10 | 0
  BMI SDS-notably low-Baseline | 0
  BMI SDS-notably low-Year 1 | 0
  BMI SDS-notably low-Year 2: number analyzed (Participants) | 14
  BMI SDS-notably low-Year 2 | 1
  BMI SDS-notably low-Year 3 | 0
  BMI SDS-notably low-Year 4 | 0
  BMI SDS-notably low-Year 5: number analyzed (Participants) | 12
  BMI SDS-notably low-Year 5 | 1
  BMI SDS-notably low-Year 6: number analyzed (Participants) | 12
  BMI SDS-notably low-Year 6 | 2
  BMI SDS-notably low-Year 7: number analyzed (Participants) | 9
  BMI SDS-notably low-Year 7 | 0
  BMI SDS-notably low-Year 8: number analyzed (Participants) | 9
  BMI SDS-notably low-Year 8 | 1
  BMI SDS-notably low-Year 9: number analyzed (Participants) | 8
  BMI SDS-notably low-Year 9 | 2
  BMI SDS-notably low-Year 10: number analyzed (Participants) | 3
  BMI SDS-notably low-Year 10 | 1
  BMI SDS-notably high-Baseline | 4
  BMI SDS-notably high-Year 1 | 1
  BMI SDS-notably high-Year 2: number analyzed (Participants) | 14
  BMI SDS-notably high-Year 2 | 1
  BMI SDS-notably high-Year 3 | 0
  BMI SDS-notably high-Year 4 | 1
  BMI SDS-notably high-Year 5: number analyzed (Participants) | 12
  BMI SDS-notably high-Year 5 | 1
  BMI SDS-notably high-Year 6: number analyzed (Participants) | 12
  BMI SDS-notably high-Year 6 | 1
  BMI SDS-notably high-Year 7: number analyzed (Participants) | 9
  BMI SDS-notably high-Year 7 | 2
  BMI SDS-notably high-Year 8: number analyzed (Participants) | 9
  BMI SDS-notably high-Year 8 | 2
  BMI SDS-notably high-Year 9: number analyzed (Participants) | 8
  BMI SDS-notably high-Year 9 | 1
  BMI SDS-notably high-Year 10: number analyzed (Participants) | 3
  BMI SDS-notably high-Year 10 | 1

3. Primary Outcome: Endocrine Laboratory Values LH and FSH in Male Participants
Description: Luteinizing hormone (LH) is a glycoprotein hormone that is co-secreted along with follicle-stimulating hormone by the gonadotrophin cells in the adenohypophysis (anterior pituitary). Untreated LH deficiency results in infertility, and if it occurs before puberty, the patient fails to develop puberty and secondary sexual characteristics. Follicle-stimulating hormone (FSH) is a hormone produced by the anterior pituitary in response to gonadotropin-releasing hormone (GnRH) from the hypothalamus. FSH plays a role in sexual development and reproduction in both males and females.
Time Frame: Annually, starting at 10-year age until 16-year age (in both studies CRAD001M2301 and CRAD001M2305)
Population: Male participants in the FAS with at least one available value of the outcome measure. In each row, the number of participants with an available value at the specified timepoint is reported.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Everolimus
Number analyzed (Participants) | 7
IU/L
  10 years age-LH: number analyzed (Participants) | 4
  10 years age-LH | 1.0 (1.47)
  10 years age-FSH: number analyzed (Participants) | 4
  10 years age-FSH | 1.5 (1.34)
  11 years age-LH: number analyzed (Participants) | 6
  11 years age-LH | 1.0 (0.77)
  11 years age-FSH: number analyzed (Participants) | 6
  11 years age-FSH | 1.7 (1.11)
  12 years age-LH | 1.8 (1.22)
  12 years age-FSH | 2.1 (0.67)
  13 years age-LH: number analyzed (Participants) | 6
  13 years age-LH | 2.4 (2.26)
  13 years age-FSH: number analyzed (Participants) | 6
  13 years age-FSH | 2.9 (1.81)
  14 years age-LH: number analyzed (Participants) | 6
  14 years age-LH | 2.9 (2.18)
  14 years age-FSH: number analyzed (Participants) | 6
  14 years age-FSH | 4.6 (4.29)
  15 years age-LH: number analyzed (Participants) | 4
  15 years age-LH | 2.5 (1.07)
  15 years age-FSH: number analyzed (Participants) | 4
  15 years age-FSH | 3.3 (0.61)
  16 years age-LH: number analyzed (Participants) | 3
  16 years age-LH | 3.5 (0.32)
  16 years age-FSH: number analyzed (Participants) | 3
  16 years age-FSH | 6.0 (3.01)

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs (any AE regardless of seriousness), AEs led to study treatment discontinuation, SAEs and SAEs led to study treatment discontinuation.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Safety Set included all pediatric patients enrolled who had at least one-post baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 14
Participants
  At least one AE | 12
  At least one SAE | 6
  AE leading to discontinuation | 0
  SAE leading to discontinuation | 0

5. Secondary Outcome: Participants Age at Menarche/Thelarche (Females) or Adrenarche (Males)
Description: Menarche is defined as the first menstrual period in a female adolescent. Menarche typically occurs between the ages of 10 and 16, with the average age of onset being 12.4 years. Thelarche is the beginning of adult breast development, marks the onset of puberty in the majority of women and occurs at a mean age of 10 years. Adrenarche refers to the time during puberty when the adrenal glands increase their production and secretion of adrenal androgens. Potential delayed puberty in girls is defined as failure to attain Tanner Stage II (for both breast development and pubic hair) by age 13, or absence of menarche by age 15 or within 5 years of attainment of Tanner Stage II. Potential delayed puberty in boys is defined as failure to attain Tanner Stage II (for both testis and pubic hair) by age 14.
Time Frame: Up to approximately 14.4 years from the first dose of everolimus in parent study CRAD001M2301 (including up to 9 years of follow-up in study CRAD001M2305)
Population: The Safety Set included all pediatric patients enrolled who had at least one-post baseline safety assessment. At each row, only participants without menarche (females), thelarche (females) and adrenarche (males) prior to start of everolimus in the parent study CRAD001M2301 are included in the analysis.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Everolimus
Number analyzed (Participants) | 14
years
  Menarche: number analyzed (Participants) | 7
  Menarche | 12.5 [11.0 to 13.6]
  Thelarche: number analyzed (Participants) | 5
  Thelarche | 10.2 [9.1 to NA] — Not estimable due to insufficient number of participants with events
  Adrenarche: number analyzed (Participants) | 7
  Adrenarche | 11.0 [10.0 to 11.6]

6. Secondary Outcome: Participants Age at Tanner Stage II, III, IV, V
Description: Tanner Staging, also known as Sexual Maturity Rating (SMR), is an objective classification system that providers use to document and track the development and sequence of secondary sex characteristics of children during puberty.
  Pubic Hair Scale
  Stages:
  II-Downy hair III-Scant terminal hair IV-Terminal hair that fills the entire triangle overlying the pubic region V-Terminal hair that extends beyond the inguinal crease onto the thigh Female Breast Development Scale
  Stages:
  II-Breast bud palpable under the areola (1st pubertal sign in females) III-Breast tissue palpable outside areola; no areolar development IV-Areola elevated above the contour of the breast, forming a "double scoop" appearance V-Areolar mound recedes into single breast contour with areolar hyperpigmentation, papillae development, and nipple protrusion Male External Genitalia Scale
  Stages:
  II- 2.5 to 3.3 cm long, 1st pubertal sign in males III- 3.4 to 4.0 cm long IV- 4.1 to 4.5 cm long V- or > 4.5 cm long
Time Frame: as for outcome 5
Population: The Full Analysis Set for sexual development (FAS Puberty) consisted of all participants enrolled in this study.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Everolimus
Number analyzed (Participants) | 15
years
  Tanner stage II-pubic hair-male: number analyzed (Participants) | 6
  Tanner stage II-pubic hair-male | 11.8 [10.2 to NA] — Not estimable due to insufficient number of participants with events
  Tanner stage II-genitalia: number analyzed (Participants) | 6
  Tanner stage II-genitalia | 11.9 [10.4 to NA] — Not estimable due to insufficient number of participants with events
  Tanner stage III-pubic hair-male: number analyzed (Participants) | 6
  Tanner stage III-pubic hair-male | 13.3 [11.3 to NA] — Not estimable due to insufficient number of participants with events
  Tanner stage III-genitalia: number analyzed (Participants) | 6
  Tanner stage III-genitalia | 12.6 [11.3 to 14.2]
  Tanner stage IV-pubic hair-male: number analyzed (Participants) | 6
  Tanner stage IV-pubic hair-male | 14.2 [11.3 to NA] — Not estimable due to insufficient number of participants with events
  Tanner stage IV-genitalia: number analyzed (Participants) | 6
  Tanner stage IV-genitalia | 14.2 [11.3 to NA] — Not estimable due to insufficient number of participants with events
  Tanner stage V-pubic hair-male: number analyzed (Participants) | 5
  Tanner stage V-pubic hair-male | 16.4 [15.3 to NA] — Not estimable due to insufficient number of participants with events
  Tanner stage V-genitalia: number analyzed (Participants) | 6
  Tanner stage V-genitalia | 16.4 [12.7 to NA] — Not estimable due to insufficient number of participants with events
  Tanner stage II-pubic hair-female: number analyzed (Participants) | 8
  Tanner stage II-pubic hair-female | 10.4 [7.3 to 11.8]
  Tanner stage II-Breast: number analyzed (Participants) | 7
  Tanner stage II-Breast | 11.5 [9.9 to 11.8]
  Tanner stage III-pubic hair-female: number analyzed (Participants) | 8
  Tanner stage III-pubic hair-female | 12.2 [10.4 to 12.8]
  Tanner stage III-Breast: number analyzed (Participants) | 7
  Tanner stage III-Breast | 12.5 [10.4 to 14.6]
  Tanner stage IV-pubic hair-female: number analyzed (Participants) | 6
  Tanner stage IV-pubic hair-female | 13.4 [11.6 to 14.5]
  Tanner stage IV-Breast: number analyzed (Participants) | 7
  Tanner stage IV-Breast | 13.8 [12.7 to 14.6]
  Tanner stage V-pubic hair-female: number analyzed (Participants) | 4
  Tanner stage V-pubic hair-female | 16.0 [13.8 to NA] — Not estimable due to insufficient number of participants with events
  Tanner stage V-Breast: number analyzed (Participants) | 2
  Tanner stage V-Breast | NA [13.8 to NA] — Not estimable due to insufficient number of participants with events

7. Secondary Outcome: TAND Checklist: Number of Participants Achieved Basic Developmental Milestones and the Age at Which Participants Achieved the Basic Developmental Milestones
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. This outcome measure assesses the TAND checklist part about basic development skills. Baseline is defined as the first available assessment on or after the enrollment date of the CRAD001M2305 study. Overall consists of all responses including baseline.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Mean (Standard Error); unit: age (months)
Arm/Group | Everolimus
Number analyzed (Participants) | 15
age (months)
  First smile-baseline | 2.9 (1.85)
  First smile-overall | 2.9 (1.85)
  Sat without support-baseline | 7.5 (3.68)
  Sat without support-overall | 7.5 (3.68)
  Walked without holding on-baseline | 16.5 (8.23)
  Walked without holding on-overall | 16.5 (8.23)
  First used single words other than "mama" or "dada"-baseline | 29.5 (24.81)
  First used single words other than "mama" or "dada"-overall | 29.5 (24.81)
  First used two words/short phrases-baseline | 33.2 (16.66)
  First used two words/short phrases-overall | 34.3 (19.77)
  Toilet trained during the day-baseline | 46.2 (31.22)
  Toilet trained during the day-overall | 51.5 (35.89)
  Toilet trained at night-baseline | 52.5 (35.60)
  Toilet trained at night-overall | 60.1 (43.23)

8. Primary Outcome: Endocrine Laboratory Values LH and FSH in Female Participants
Description: as for outcome 3
Time Frame: Annually, starting at 10-year age until 16-year age (in both studies CRAD001M2301 and CRAD001M2305)
Population: Female participants in the FAS with at least one available value of the outcome measure. In each row, the number of participants with an available value at the specified timepoint is reported.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Everolimus
Number analyzed (Participants) | 8
IU/L
  10 years age-LH: number analyzed (Participants) | 2
  10 years age-LH | 5.1 (3.89)
  10 years age-FSH: number analyzed (Participants) | 2
  10 years age-FSH | 3.4 (2.68)
  11 years age-LH: number analyzed (Participants) | 7
  11 years age-LH | 3.2 (2.47)
  11 years age-FSH: number analyzed (Participants) | 7
  11 years age-FSH | 3.5 (1.61)
  12 years age-LH: number analyzed (Participants) | 7
  12 years age-LH | 7.8 (6.73)
  12 years age-FSH: number analyzed (Participants) | 7
  12 years age-FSH | 5.6 (2.43)
  13 years age-LH: number analyzed (Participants) | 5
  13 years age-LH | 4.4 (3.08)
  13 years age-FSH: number analyzed (Participants) | 5
  13 years age-FSH | 5.0 (0.80)
  14 years age-LH: number analyzed (Participants) | 6
  14 years age-LH | 5.3 (6.97)
  14 years age-FSH: number analyzed (Participants) | 6
  14 years age-FSH | 2.6 (2.05)
  15 years age-LH: number analyzed (Participants) | 4
  15 years age-LH | 7.5 (10.96)
  15 years age-FSH: number analyzed (Participants) | 4
  15 years age-FSH | 2.5 (2.28)
  16 years age-LH: number analyzed (Participants) | 4
  16 years age-LH | 3.7 (2.69)
  16 years age-FSH: number analyzed (Participants) | 4
  16 years age-FSH | 2.8 (2.05)

9. Primary Outcome: Endocrine Laboratory Values of Testosterone in Male Participants
Description: Testosterone is the primary male hormone responsible for regulating sex differentiation, producing male sex characteristics, spermatogenesis, and fertility.
Time Frame: Annually, starting at 10-year age until 16-year age (in both studies CRAD001M2301 and CRAD001M2305)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Everolimus
Number analyzed (Participants) | 7
nmol/L
  10 years age: number analyzed (Participants) | 4
  10 years age | 0.7 (1.17)
  11 years age: number analyzed (Participants) | 6
  11 years age | 2.5 (4.60)
  12 years age | 3.8 (4.29)
  13 years age: number analyzed (Participants) | 6
  13 years age | 4.3 (4.04)
  14 years age: number analyzed (Participants) | 6
  14 years age | 7.2 (4.34)
  15 years age: number analyzed (Participants) | 4
  15 years age | 12.9 (6.28)
  16 years age: number analyzed (Participants) | 3
  16 years age | 15.5 (3.93)

10. Primary Outcome: Endocrine Laboratory Values of Estrogen in Female Participants
Description: Estrogen is a steroid hormone associated with the female reproductive organs and is responsible for developing female sexual characteristics.
Time Frame: Annually, starting at 10-year age until 16-year age (in both studies CRAD001M2301 and CRAD001M2305)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Everolimus
Number analyzed (Participants) | 8
ng/L
  10 years age: number analyzed (Participants) | 1
  10 years age | 139.8
  11 years age: number analyzed (Participants) | 4
  11 years age | 80.5 (119.22)
  12 years age: number analyzed (Participants) | 3
  12 years age | 43.7 (41.26)
  13 years age: number analyzed (Participants) | 2
  13 years age | 50.0 (7.07)
  14 years age: number analyzed (Participants) | 2
  14 years age | 139.0 (141.42)
  15 years age: number analyzed (Participants) | 4
  15 years age | 47.7 (48.89)
  16 years age: number analyzed (Participants) | 4
  16 years age | 149.7 (128.21)

11. Secondary Outcome: TAND Checklist: Number of Participants With Behavioral Disorders
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas.
  Behavioral level- This level refers to any observed behaviors that may cause concern to the individual. Behavioral presentations include anxiety, depressed mood, aggressive behaviors, temper tantrums, attention-related behaviors (such as difficulty concentrating, hyperactivity, impulsivity), social, and communication-related behaviors (such as speech and language delays, poor eye contact, difficulties in relationships with peers, repetitive behaviors), self-injurious behaviors, and eating or sleep difficulties.
  Baseline is defined as the first available assessment on or after the enrollment date of the CRAD001M2305 study. Overall consists of all responses including baseline.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Anxiety-baseline | 12
  Anxiety-overall | 13
  Depressed mood-baseline | 6
  Depressed mood-overall | 8
  Extreme shyness-baseline | 5
  Extreme shyness-overall | 7
  Mood swings-baseline | 10
  Mood swings-overall | 12
  Aggressive outbursts-baseline | 7
  Aggressive outbursts-overall | 11
  Temper Tantrums-baseline | 9
  Temper Tantrums-overall | 12
  Self-injury, such as hitting self, biting self, scratching self-baseline | 3
  Self-injury, such as hitting self, biting self, scratching self-overall | 5
  Absent or delayed onset of language to communicate-baseline | 11
  Absent or delayed onset of language to communicate-overall | 12
  Repeating words or phrases over and over again-baseline | 9
  Repeating words or phrases over and over again-overall | 12
  Poor eye contact-baseline | 6
  Poor eye contact-overall | 8
  Difficulties getting on with other people of similar age-baseline | 9
  Difficulties getting on with other people of similar age-overall | 10
  Repetitive behaviours, such as doing the same thing over and over again-baseline | 9
  Repetitive behaviours, such as doing the same thing over and over again-overall | 11
  Very rigid or inflexible about how to do things or not liking change in routines-baseline | 8
  Very rigid or inflexible about how to do things or not liking change in routines-overall | 11
  Overactivity/hyperactivity, such as being constantly on the go-baseline | 8
  Overactivity/hyperactivity, such as being constantly on the go-overall | 9
  Difficulty paying attention or concentrating-baseline | 13
  Difficulty paying attention or concentrating-overall | 15
  Restlessness or fidgetiness, such as wriggling or squirming-baseline | 13
  Restlessness or fidgetiness, such as wriggling or squirming-overall | 14
  Impulsivity, such as butting in, not waiting turn-baseline | 10
  Impulsivity, such as butting in, not waiting turn-overall | 12
  Difficulties with eating, such as eating too much, too little, unusual things-baseline | 5
  Difficulties with eating, such as eating too much, too little, unusual things-overall | 8
  Sleep difficulties, such as with falling asleep or waking-baseline | 6
  Sleep difficulties, such as with falling asleep or waking-overall | 8

12. Secondary Outcome: TAND Checklist - Number of Participants With Psychiatric Disorders
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. For psychiatric disorders some behaviors of concern are examined and evaluated in the context of the individual's overall developmental level and in terms of their biological, psychological, and social profile. Baseline is defined as the first available assessment on or after the enrollment date of the CRAD001M2305 study. Overall consists of all responses including baseline.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Autism Spectrum Disorder (ASD), including autism, Asperger's-baseline | 4
  Autism Spectrum Disorder (ASD), including autism, Asperger's-overall | 7
  Attention Deficit Hyperactivity Disorder (ADHD)-baseline | 5
  Attention Deficit Hyperactivity Disorder (ADHD)-overall | 9
  Anxiety Disorder, including as panic, phobia, separation anxiety disorder-baseline | 4
  Anxiety Disorder, including as panic, phobia, separation anxiety disorder-overall | 7
  Depressive Disorder-baseline | 0
  Depressive Disorder-overall | 0
  Obsessive Compulsive Disorder-baseline | 2
  Obsessive Compulsive Disorder-overall | 2
  Psychotic Disorder, including schizophrenia-baseline | 0
  Psychotic Disorder, including schizophrenia-overall | 0

13. Secondary Outcome: TAND Checklist - Number of Participants With Scholastic Issues
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. At academic level, it is described the specific learning disorders associated with school performance, such as reading, writing, mathematics, and spelling. Baseline is defined as the first available assessment on or after the enrollment date of the CRAD001M2305 study. Overall consists of all responses including baseline.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Reading-baseline | 12
  Reading-overall | 14
  Writing-baseline | 12
  Writing-overall | 14
  Spelling-baseline | 12
  Spelling-overall | 14
  Mathematics-baseline | 12
  Mathematics-overall | 14

14. Secondary Outcome: TAND Checklist: Number of Participants With Difficulty in Specific Brain Skills
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. Neuropsychological evaluations are used to describe the strengths and weaknesses of brain referenced systems used for learning, thinking, and behavior regulation. Baseline is defined as the first available assessment on or after the enrollment date of the CRAD001M2305 study. Overall consists of all responses including baseline.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Memory-baseline | 7
  Memory-overall | 12
  Attention-baseline | 12
  Attention-overall | 14
  Dual-tasking/ Multi-tasking-baseline | 12
  Dual-tasking/ Multi-tasking-overall | 14
  Visuo-spatial tasks-baseline | 8
  Visuo-spatial tasks-overall | 13
  Executive skills-baseline | 10
  Executive skills-overall | 15
  Getting disoriented-baseline | 7
  Getting disoriented-overall | 12

15. Secondary Outcome: TAND Checklist - Number of Participants With Psychological Issues
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. At psychosocial level it is considered important determinants of quality of life, such as self-esteem, family functioning, parental stress, and relationship difficulties. All these are markers of resilience and burden of care, and all the psychosocial factors may be amenable to intervention and support. Baseline is defined as the first available assessment on or after the enrollment date of the CRAD001M2305 study. Overall consists of all responses including baseline.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Low self-esteem-baseline | 2
  Low self-esteem-overall | 6
  Very high levels of stress in families, for instance between siblings-baseline | 6
  Very high levels of stress in families, for instance between siblings-overall | 8
  Very high levels of stress between parents leading to significant relationship difficulties-baseline | 5
  Very high levels of stress between parents leading to significant relationship difficulties-overall | 7

16. Secondary Outcome: TAND Checklist - Number of Participants With Varied Levels of Language Skills
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. Neuropsychological evaluations are used to describe the strengths and weaknesses of brain referenced systems used for learning, thinking, and behavior regulation. These include language skills (including non-verbal, simple language, fluence of language). All the responses are categorical in nature from the TAND Checklist. The frequency of (baseline and) worst-post baseline is summarized.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Non-verbal | 2
  Simple language | 6
  Fluent | 4
  Missing | 3

17. Secondary Outcome: TAND Checklist - Number of Participants With Different Levels of Physical Dependency
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. This outcome measure assesses the TAND checklist part about physical dependency. All the responses are categorical in nature from the TAND Checklist. The frequency of (baseline and) worst-post baseline is summarized.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Dependent on others | 4
  Some self-care skills | 7
  Independent | 1
  Missing | 3

18. Secondary Outcome: TAND Checklist: Number of Participants With Different Levels of Mobility
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. This outcome measure assesses the TAND checklist part about mobility. All the responses are categorical in nature from the TAND Checklist. The frequency of (baseline and) worst-post baseline is summarized.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Wheelchair | 1
  Needs significant support | 1
  Some difficulty | 0
  Completely mobile | 10
  Missing | 3

19. Secondary Outcome: TAND Checklist: Number of Participants With Different Levels of Intelligence Quotient
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. At intellectual level, it is described the intellectual developmental abilities of an individual in comparison with others of the same chronological age. All the responses are categorical in nature from the TAND Checklist. The frequency of (baseline and) worst-post baseline is summarized.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Normal Intellectual Ability (IQ > 80) | 2
  Borderline Intellectual Ability (IQ 70-80) | 2
  Mild Intellectual Disability (IQ 50-69) | 1
  Moderate Intellectual Disability (IQ 35-49) | 5
  Severe Intellectual Disability (IQ 21-34) | 0
  Profound Intellectual Disability (IQ <20) | 1
  Missing | 4

20. Secondary Outcome: TAND Checklist: Number of Participants With Different Levels of Intellectual Ability
Description: Tuberous Sclerosis Complex (TSC) is associated with a range of neuropsychiatric disorders which refers to as TAND (TSC-Associated-Neuropsychiatric-Disorders). A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas. At intellectual level, it is described the intellectual developmental abilities of an individual to identify their overall functional and adaptive behaviors in comparison with others of the same chronological age. This level is the combination of formal measures of intellectual ability (such as IQ-type tests) and evaluation of adaptive behaviors (such as self-care, daily living skills, communication, and social abilities in daily life). All the responses are categorical in nature from the TAND Checklist. The frequency of (baseline and) worst-post baseline is summarized.
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Population: The Full Analysis Set (FAS) consisted of all participants enrolled in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 15
Participants
  Normal Intellectual Ability | 1
  Mild-Moderate Intellectual Disability | 8
  Severe - Profound Intellectual Disability | 3
  Missing | 3

ADVERSE EVENTS:
Time Frame: From enrollment in study CRAD001M2305 until end of study, up to approximately 9 years.
Description: Adverse events are assessed in the Safety Set. The Safety Set included all pediatric patients enrolled who had at least one-post baseline safety assessment.
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=14)
Drowning (General disorders) | 1
Pyrexia (General disorders) | 2
Arthritis infective (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Near drowning (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 2
Status epilepticus (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=14)
Anaemia (Blood and lymphatic system disorders) | 3
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Right ventricular dilatation (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Periorbital swelling (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Gingival hypertrophy (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Microsomia (General disorders) | 1
Pyrexia (General disorders) | 6
Seasonal allergy (Immune system disorders) | 3
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Croup infectious (Infections and infestations) | 1
Ear infection (Infections and infestations) | 4
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 4
Otitis media (Infections and infestations) | 2
Pharyngitis streptococcal (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Cardiac murmur (Investigations) | 1
Cutibacterium test positive (Investigations) | 1
SARS-CoV-2 test negative (Investigations) | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Head discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 4
Vasogenic cerebral oedema (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 3
Attention deficit hyperactivity disorder (Psychiatric disorders) | 2
Euphoric mood (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Central sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 3

LIMITATIONS AND CAVEATS:
It was anticipated that maximum of 50 patients who have participated in Study M2301 would be eligible to enter Study M2305 if they consent to participate. However, only 15 patients were enrolled into this study, due to delays in study start-up at country level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-08-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT02338609/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT02338609/SAP_001.pdf